CLINICAL TRIAL: NCT02044601
Title: Phase I/II Trial Using a Biomarker-Integrated Approach of Targeted Therapy for Lung Cancer Elimination Plus External Beam Radiation Therapy (BATTLE-XRT)
Brief Title: Biomarker-Integrated Approach of Targeted Therapy for Lung Cancer Elimination Plus External Beam Radiation Therapy (BATTLE-XRT)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0556
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; NSCLC; Squamous cell carcinoma of the lung; Adenocarcinoma of the lung; Radiation therapy; Proton therapy; XRT; Carboplatin; Paraplatin; Paclitaxel; Taxol; Onartuzumab; Erlotinib; Erlotinib hydrochloride; OSI-774; CP358774; Tarceva
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — onartuzumab; Erlotinib Hydrochloride; Paclitaxel; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiation + Onartuzumab (Experimental): Participants with wild-type EGFR mutation to be randomized, and may receive this regimen.
  Phase I: Starting dose of Onartuzumab 10 mg/kg by vein on Day 1 of each 3 week cycle. Paclitaxel 45 mg/m2 by vein once a week throughout radiation for 7 weeks. Carboplatin AUC 2 by vein once a week throughout radiation for 7 weeks. Radiation therapy at 66 Gy in 33 fractions delivered 5 days a week for 7 weeks, or proton therapy delivered at biological equivalent to 66 Gy (RBE) (RBE = 1.1) in 33 fractions 5 days a week for 7 weeks.
  Phase II: Same regimen as in Phase I, but starting dose of Onartuzumab is maximum tolerated dose from Phase I.
  Interventions: Drug: Onartuzumab; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiation Therapy
- Chemoradiation + Erlotinib + Onartuzumab (Experimental): Participants with EGFR mutation to receive this regimen. Participants with wild-type EGFR mutation to be randomized, and may receive this regimen.
  Phase I: Erlotinib 150 mg by mouth every day throughout radiation, except for chemotherapy day. Starting dose of Onartuzumab 10 mg/kg by vein on Day 1 of each 3 week cycle. Paclitaxel 45 mg/m2 by vein once a week throughout radiation for 7 weeks. Carboplatin AUC 2 by vein once a week throughout radiation for 7 weeks. Radiation therapy at 66 Gy in 33 fractions delivered 5 days a week for 7 weeks, or proton therapy delivered at biological equivalent to 66 Gy (RBE) (RBE = 1.1) in 33 fractions 5 days a week for 7 weeks.
  Phase II: Same regimen as in Phase I, but starting dose of Onartuzumab is maximum tolerated dose from Phase I.
  Interventions: Drug: Onartuzumab; Drug: Erlotinib; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Onartuzumab — Phase I: Starting dose of Onartuzumab 10 mg/kg by vein on Day 1 of each 3 week cycle.
  Phase II: Maximum tolerated dose from Phase I.
Drug: Erlotinib — Phase I and II: 150 mg by mouth every day throughout radiation, except for chemotherapy day.
  Other Names: Erlotinib Hydrochloride; OSI-774; CP358774; Tarveva
  Arms: Chemoradiation + Erlotinib + Onartuzumab
Drug: Paclitaxel — Phase I and II: 45 mg/m2 by vein once a week throughout radiation for 7 weeks.
  Other Names: Taxol
Drug: Carboplatin — Phase I and II: AUC 2 by vein once a week throughout radiation for 7 weeks.
  Other Names: Paraplatin
Radiation: Radiation Therapy — Phase I and II: Radiation therapy at 66 Gy in 33 fractions delivered 5 days a week for 7 weeks, or proton therapy delivered at biological equivalent to 66 Gy (RBE) (RBE = 1.1) in 33 fractions 5 days a week for 7 weeks.
  Other Names: XRT

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of onartuzumab that can be given with erlotinib and standard chemoradiation (paclitaxel and carboplatin) to patients with NSCLC.

The goal of Phase II is to learn if onartuzumab plus erlotinib and chemoradiation can help to control NSCLC. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study and you have an EGFR mutation, you will be enrolled in Arm A. If you have the wild-type EGFR, you will be randomly assigned (as in the flip of a coin) to either Arm B or C. You will have an equal chance of being enrolled in either arm.

* If you are in Arm A, you will receive standard chemoradiation, erlotinib, and onartuzumab.
* If you are in Arm B, you will receive standard chemoradiation, erlotinib, and onartuzumab.
* If you are in Arm C, you will receive standard chemoradiation and onartuzumab only.

If you are assigned to Arm A or B, you will receive standard chemoradiation, erlotinib, and onartuzumab. You will be assigned to a dose level of onartuzumab based on when you join this study. After the first dose level of onartuzumab is given, you will be watched for 2 weeks after the end of radiation treatment to check for any serious side effects at that dose level. If any participants in this first group have intolerable side effects, a lower dose combination of the study drugs may be tested. Once the highest tolerable dose is found, extra participants will receive onartuzumab at that dose level.

All participants in Arms A and B will receive the same dose level of erlotinib.

Study Drug Administration:

All participants will receive onartuzumab by vein on Day 1 of each 3-week cycle. The first infusion should be given over about 60 minutes. If the infusion is tolerated, other doses will be given over about 30 minutes.

You will receive paclitaxel and carboplatin by vein over about 6 hours 1 time a week for 7 weeks. You will receive a separate consent form for chemoradiation, which will describe the procedure and risks in more detail.

If you are taking erlotinib, it should be taken by mouth with about 1 cup of water. You should take erlotinib at about the same time every day, at least 1 hour before a meal and at least 2 hours after a meal.

Study Visits:

One (1) time each week:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests. If you are taking Coumadin or a similar drug, this blood will also be used to check how well your blood clots.

Length of Study:

You may continue taking onartuzumab until you complete radiation therapy. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over 4 years after your last dose of study drug.

Follow-Up:

You will have follow-up visits around 30 days after your last dose of study drug, every 3 months for 2 years, and then every 4 months for the next 2 years. During these visits:

* You will have a physical exam.
* You will have a CT or PET scan to check the status of the disease.
* If you are taking Coumadin or a similar drug, blood (about 2 teaspoons) will be drawn to check how well your blood clots.

You will be called about every 4 weeks and asked how you are doing for as long as your doctor thinks it is needed.

This is an investigational study. Onartuzumab is not FDA approved or commercially available. It is currently being used for research purposes only. Erlotinib, carboplatin, and paclitaxel are all FDA approved and commercially available for the treatment of NSCLC, but their use in this study is investigational. Radiation therapy is delivered using FDA-approved and commercially available methods. The study doctor can explain how the study drugs are designed to work.

Up to 90 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented NSCLC, including squamous cell carcinoma, adenocarcinoma (including bronchoalveolar cell), and large cell anaplastic carcinoma (including giant and clear cell carcinomas) and poorly differentiated (not otherwise specified, NOS) non-small cell lung cancer; totally resected tumors are excluded. Patients should have tumor tissue for biomarker testing if available. Archival samples may be used. Patients without tissue for biomarker testing may be enrolled at the discretion of the investigator. The determination of MET status should be done by a pathologist who is trained in using the SP44 antibody with the Ventana platform and using the Ventana/Genentech algorithm.
2. Patients with T1or T2 disease with N2 or T3N1-2 disease (Stage IIIA) are eligible if they are deemed inoperable. Patients with T4 with any N or any T with N2 or N3 disease are eligible if unresectable. Patients may have limited stage M1 disease, with a maximum of 3 metastatic sites (including the single brain mets) only if the other sites are to be treated with definitive intent, unless they are no longer clinically present secondary to induction chemotherapy. Treatment to the other sites can be delivered prior to or after this trial. Measurable disease is required. See Response Evaluation Criteria in Solid Tumors (RECIST) definitions of measurable disease.
3. Patients must be >/=18 years of age.
4. Patients with Zubrod performance status 0-2.
5. Adequate hematologic function defined as: ANC >/= 1,500/mm3, platelets >/= 100,000/mm3, and hemoglobin >/= 9 g/dL (prior to transfusions); adequate hepatic function defined as: total bilirubin </= 1.5 mg/dl, SGOT or SGPT </= 3 x ULN, adequate renal function defined as a serum creatinine level </= 2.0 mg/dl, alkaline phosphatase </= 2.5 x ULN, glucose </= 2 x ULN.
6. FEV1 with >/= 1000 cc.
7. Patients with a pleural effusion that is a transudate, cytologically negative and nonbloody are eligible if the radiation oncologists feel the tumor can still be encompassed within a reasonable field of radiotherapy. If a pleural effusion can be seen on the chest computed tomography (CT) but not on chest x-ray (CXR) and is too small to tap, the patient is eligible.
8. If patients had exploratory thoracotomy, they must have recovered from the procedure (</= grade 1 or baseline). Exploratory Thoracotomy and beginning of treatment should be within one month.
9. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for four weeks after completion of treatment.
10. For women of childbearing potential, a urine or blood pregnancy test must be performed within 48 hours prior to the start of protocol treatment.
11. Prior induction chemotherapy will be allowed, as is prior target therapy. Patients with progression on an EGFR targeting agent will also be allowed, but stratified between the two arms.
12. Patients must sign a study-specific consent form prior to study entry.

Exclusion Criteria:

1. Active pulmonary infection not responsive to conventional antibiotics
2. History of interstitial lung disease.
3. History of severe chronic obstructive pulmonary disease (COPD) requiring >/= 3 hospitalizations over the past year.
4. Significant history of cardiac disease, i.e., uncontrolled hypertension (i.e. can't reduce blood pressure (BP) below a systolic of 160 or diastolic of 100), unstable angina, uncompensated congestive heart failure, myocardial infarction within the past 2 months, or cardiac ventricular arrhythmias requiring medication.
5. Patients with > grade 3 neuropathy.
6. Evidence of life threatening disease resulting in a life expectancy of less than 3 months.
7. Women who are pregnant or breast feeding, as treatment involves unforeseeable risks to the participant, embryo, fetus, or nursing infant; women with a positive pregnancy test on enrollment or prior to study drug administration.
8. Women of childbearing potential and male participants who are unwilling or unable to use an acceptable method of contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for four weeks after completion of treatment or those who are using a prohibited contraceptive method (methods with unknown efficacy).
9. Patients who currently are participating in other clinical trials and/or who have participated in other clinical trials (These patient may be enrolled but radiation must not start within 15 days of any previous experiment therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Onartuzumab with Chemoradiation Therapy and Erlotinib | 6 months
  Maximum tolerated dose measured by the number and percent of patients experiencing dose-limiting toxicity (DLT). DLT defined as grade 3 or worse non-hematological toxicities or grade 4 or worse hematological toxicities (including all toxicities attributed to chemoradiation occurring up to 14 days of the end of radiation therapy).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Progression-free survival defined by 6-month progression free survival. Response is taken to be complete response (CR) or partial response (PR) using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org